CLINICAL TRIAL: NCT06783062
Title: Activation Failure of Knee Extensors After Anterior Cruciate Ligament Rupture Depending on the Contraction Mode
Acronym: QUADFAIL
Status: Not yet recruiting | Type: Observational
Sponsor: La Tour Hospital (Other)
Collaborators: Toulouse NeuroImaging Center (ToNIC - UMR 1214 Inserm/UPS) (Unknown)
Responsible Party: Principal Investigator, Simon Barrué-Belou, Physiotherapist PhD., in charge of Biomechanics, La Tour Hospital
Other Study IDs: 2024-01580
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture; Activation Failure; Contraction Mode
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control
- ACL - rehabilitation
- ACL - surgery + rehabilitation

SUMMARY:
The primary objective of the study is to evaluate the impact of ACL injury and ACL reconstruction on voluntary activation during maximal voluntary contraction (measured by neurophysiological parameters) according to the contraction mode.

The goal is to provide elements of knowledge to clinicians about the mechanisms of the activation failure depending on contraction mode, but also the resulting adapted clinical recommendations for conducting rehabilitation, and particularly for the use of different contraction modes.

The main hypothesis is that activation failure is not equal according to the contraction mode during maximal voluntary contractions and neurophysiological parameters will be decreased in comparison with non-injured subjects.

Secondary objectives are:

* To analyze the evolution of neurophysiological parameters between sessions interspaced by several months according to the contraction mode.
* To observe this time evolution depending on the treatment strategy chosen: rehabilitation or surgery plus rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

A. ACL-injured groups (surgically or conservatively treated):

1. Age between 18 and 50 years
2. Free, informed consent signed by the participant and the investigator.
3. Session 1: Delay of 2 to 6 weeks after injury, with a quiet knee (range of motion 110- 0°, minimal effusion, maximal contraction pain ≤ 2/10)
4. Session 2: Duration of 36 to 42 weeks after injury, with a quiet knee (range of motion 110-0°, minimal effusion, maximal contraction pain ≤ 2/10)
5. Independent person (Unprotected: under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision)

B. ControlGroup:

1. Age between 18 and 50 years
2. Free, informed consent signed by the participant and the investigator.
3. Sport practitioners: at least once per week practicing activities like collective sports, racket sports, combat sports, skiing, or on-loading activities with changing of directions.
4. Independent person (Unprotected: under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision)

Exclusion Criteria:

* 1. Subjects fitted with an implanted electronic device such as a cardiac pacemaker 2. Professional athlete 3. Pregnant women 4. Subject with systemic pathology or treatment affecting the musculoskeletal system 5. Subject with a history of neurological pathology or traumatic pathology, or pathology that required orthopedic treatment and/or surgery of the knee, hip and/or lumbar spine 6. Contraindication to isokinetic testing: incapacitating pain, evolving pathological process, non- healed fracture, unbalanced cardiovascular pathology (angina pectoris, arterial hypertension) 7. Contralateral knee injury 8. Subject inability to follow procedures or insufficient knowledge of project language 9. Data acquisition issue or injury during testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will comprise both male and female subjects, divided into three groups. The first group will consist of 20 subjects with isolated (only ACL rupture) or non-isolated ACL rupture (rupture associated with other knee lesion), treated with rehabilitation. The second group will include 20 subjects with ACL rupture, treated with surgery and rehabilitation. A third control group will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Voluntary Activation Level | Between 2 and 6 weeks after ACL rupture

SECONDARY OUTCOMES:
Maximal voluntary torque | between 2 to 6 weeks after ACL rupture
EMG activity of vastus lateralis, vastus medialis and rectus femoris | between 2 to 6 weeks after ACL rupture
  Quantified with root mean square (RMS), normalized to the maximal M-wave
Voluntary Activation Level | Around 9 months after ACL rupture
Maximal voluntary torque | Around 9 months after ACL rupture
EMG activity of vastus lateralis, vastus medialis and rectus femoris | Around 9 months after ACL rupture

IPD SHARING:
Plan to Share IPD: Undecided